CLINICAL TRIAL: NCT00940134
Title: INGEAR-1: Effects of INtravenous Infusions of PYY3-36 and GLP-1, as Monoinfusion and in Combination, on ad Libitum Energy Intake, Appetite Sensation, and Energy Expenditure in Healthy Obese Subjects.
Brief Title: Effects of Intravenous Infusions of Gut Hormones on Appetite and Metabolism.
Acronym: INGEAR-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, AAstrup, Professor, MD, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B262
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Obesity
Keywords: obesity; energy expenditure; incretins; appetite regulation; GLP-1; PYY; ad libitum energy intake
MeSH Terms: conditions — Obesity | interventions — peptide YY (3-36); Glucagon-Like Peptide 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- placebo (Placebo Comparator): Study participants will receive a 3 hour IV infusion of saline while fasting.
  Interventions: Biological: saline infusion
- PYY3-36 + GLP-1 (Experimental): Study participants will receive a 3 hour IV infusion of (GLP-1 + PYY3-36) while fasting.
  Interventions: Biological: PYY 3-36; Biological: GLP-1
- GLP-1 (Active Comparator): Study participants will receive a 3 hour IV infusion of PYY3-36 while fasting.
  Interventions: Biological: GLP-1
- PYY3-36 (Active Comparator): Study participants will receive a 3 hour IV infusion of PYY3-36 while fasting.
  Interventions: Biological: PYY 3-36

INTERVENTIONS:
Biological: PYY 3-36 — 0.8 pmol/kg/min x 3 hours
  Arms: PYY3-36; PYY3-36 + GLP-1
Biological: GLP-1 — 1.0 pmol/kg/min x 3 hours
  Arms: GLP-1; PYY3-36 + GLP-1
Biological: saline infusion — saline infusion x 3 hours
  Arms: placebo

SUMMARY:
The purpose of this study is to investigate the effects of intravenous infusion of two gastrointestinal hormones, PYY3-36 and GLP-1, alone and in combination, on appetite in healthy obese men. The investigators hypothesize that an intravenous infusion of each hormone alone will decrease food intake at a buffet meal and decrease appetite, and that in combination, there will be a greater decrease in food intake and appetite compared to each hormone alone.

ELIGIBILITY:
Inclusion Criteria:

* Men age 18-50 years
* BMI ≥30
* healthy

Exclusion Criteria:

* Diabetes mellitus
* psychological illness
* on special diets (eg vegetarian, Atkins)
* weight change of >3kg within the 2 months prior to screening
* Hypothalamic or genetic aetiology of obesity
* diagnosed cancer
* chronic illness or disease
* Eating disorder (anorexia or bulimia)
* smoking
* substance abuse
* Use of any prescription or over the counter medication that can affect metabolism
* Excessive intake of alcohol (>7 drinks/week)
* Excessive intake of caffeine (>300 mg/day)
* High level of physical activity (>10 hours/week)
* Lack of desire or willingness to take part in and follow study protocol

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Ad libitum energy intake | Immediately following 3h IV infusion

SECONDARY OUTCOMES:
Energy expenditure (ventilated hood technique). | During 3h IV infusion
Changes in levels of glucose, insulin, C peptide, GIP, leptin, ghrelin, adiponectin, cholecystokinin | Prior to, and 15, 30, 60, 90, 120, 180 mins during IV infusion
Appetite sensation by visual analog scale | Every 30 minutes during 3h IV infusion
Gastric emptying (paracetamol) | At time=15, 30, 60, 90, 120, 180 mins during IV infusion

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaj T Gregersen, MSc, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Human Nutrition, Faculty of Life Sciences, University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Schmidt JB, Gregersen NT, Pedersen SD, Arentoft JL, Ritz C, Schwartz TW, Holst JJ, Astrup A, Sjodin A. Effects of PYY3-36 and GLP-1 on energy intake, energy expenditure, and appetite in overweight men. Am J Physiol Endocrinol Metab. 2014 Jun 1;306(11):E1248-56. doi: 10.1152/ajpendo.00569.2013. Epub 2014 Apr 15. PMID 24735885